CLINICAL TRIAL: NCT05849259
Title: Caring for Caregivers and People Living With Dementia Under Home-Based Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Retirement Research Foundation (Other)
Responsible Party: Principal Investigator, Christine S. Ritchie, MD, MPH, Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022P003057
Record Dates: First submitted 2023-04-07; First posted 2023-05-08 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Dementia; Quality of Life; Caregiver Stress
MeSH Terms: conditions — Dementia; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: A live open-pilot trial will be conducted of the HBPC Dementia Care Quality at Home intervention in two HBPC practices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dementia Care Quality at Home (Experimental): Caregivers across two HBPC practices receive the Dementia Care Quality at Home intervention.
  Interventions: Other: Dementia Care Quality at Home

INTERVENTIONS:
Other: Dementia Care Quality at Home — Each of the two HBPC practices will identify at least two trained Dementia Care Quality at Home Champions who will be trained in the intervention comprised of 1) a standardized assessment tool to assess PLWD and caregiver needs; 2) six modules created to optimize the well-being of the PLWD and their caregiver; and 3) regular team-based review of persons participating in the program to address care challenges and a team-based case conference approach to solve these challenges.

SUMMARY:
The goal of this clinical trial is to develop a dementia care intervention for persons receiving home-based primary care (HBPC) and living with dementia (PLWD) and their caregivers, and test the feasibility of implementing the intervention in HBPC practices to ultimately improve outcomes of PLWD and their caregivers.

The main aims are to:

* Develop and refine HBPC Dementia Care Quality at Home
* Establish feasibility (primary outcome), acceptability, and fidelity of HBPC Dementia Care Quality at Home through an open-pilot trial involving two HBPC practices. Trained clinicians and staff at two HBPC practices will implement the intervention

Relevant stakeholders (caregivers of PLWD, and HBPC clinicians and staff) will participate in qualitative focus groups to provide feedback on the intervention.

DETAILED DESCRIPTION:
The overarching goal of this project is to develop a dementia care intervention for PLWD and their caregivers, Dementia Care Quality at Home, and test the feasibility of implementing the intervention in two HBPC practices to ultimately improve outcomes of PLWD and their caregivers.

The investigators will evaluate the feasibility, acceptability, and fidelity in implementing HBPC Dementia Care Quality at Home in two practices for persons living with dementia and their caregivers through an open pilot. Hypothesis: HBPC Dementia Care Quality at Home will meet benchmarks of feasibility, acceptability, and fidelity by the HBPC practices implementing it and by caregivers of PLWD who experience the intervention. The investigators will assess feasibility of caregivers of PLWD to engage with the intervention, the acceptability of the intervention to caregivers, and the impact of the intervention on caregiver well-being by surveying caregivers at the conclusion of the pilot. In addition, the investigators will assess feasibility, acceptability, and fidelity of the intervention in the practices.

ELIGIBILITY:
Inclusion Criteria:

Caregiver participants will:

* be adults (18 years or older)
* have English fluency and literacy
* live in the United States
* live with and care for an individual with Alzheimer's Disease and Alzheimer's Disease Related Dementias (ADRD)
* anticipate providing care for the next 6 months
* provide an average 4 hours of supervision or direct assistance per day for the care recipient and
* have been identified by the practice as experiencing caregiver stress.

Staff participants will:

* be 18 years or older
* have English fluency and literacy and live in the United States and
* be part of a HBPC primary care program or closely connected to the practice.

Exclusion Criteria:

* Participants under the age 18.
* Participants who have no English fluency and literacy and do not live in the United States.
* For caregiver participants, not caring for and living with a patient that is part of a HBPC primary care program or closely connected to the practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine S Ritchie, MD, MSPH, Principal Investigator — Massachusetts General Hospital; Bruce Leff, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Queens Medical Center, Honolulu, Hawaii
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leff B, Ritchie C, Freeland DG, Jamshed N, Major A, Gallopyn N, Sharieff S, Taylor J, Yudin JA, Sheehan OC. The National Home-Based Primary Care Learning Network: A Practice-Based Quality Improvement and Research Network. J Am Med Dir Assoc. 2022 Aug;23(8):1424-1426. doi: 10.1016/j.jamda.2022.02.017. Epub 2022 Mar 26. PMID 35351444
- [Background] Foakes G, Hurt C, Lehner JL, Tinsley H, Valentine J, Doede DD, Ritchie C, Leff B. Using Registry Data to Support National Quality Forum Endorsement of Quality Measures for Home-Based Medical Care. Am J Med Qual. 2021 Nov-Dec 01;36(6):402-407. doi: 10.1097/01.JMQ.0000735496.32223.40. PMID 33990472
- [Background] Yang M, Pajewski N, Espeland M, Easterling D, Williamson JD. Modifiable risk factors for homebound progression among those with and without dementia in a longitudinal survey of community-dwelling older adults. BMC Geriatr. 2021 Oct 18;21(1):561. doi: 10.1186/s12877-021-02506-1. PMID 34663232
- [Background] Reckrey JM, Yang M, Kinosian B, Bollens-Lund E, Leff B, Ritchie C, Ornstein K. Receipt Of Home-Based Medical Care Among Older Beneficiaries Enrolled In Fee-For-Service Medicare. Health Aff (Millwood). 2020 Aug;39(8):1289-1296. doi: 10.1377/hlthaff.2019.01537. PMID 32744949
- [Background] Ornstein KA, Leff B, Covinsky KE, Ritchie CS, Federman AD, Roberts L, Kelley AS, Siu AL, Szanton SL. Epidemiology of the Homebound Population in the United States. JAMA Intern Med. 2015 Jul;175(7):1180-6. doi: 10.1001/jamainternmed.2015.1849. PMID 26010119
- [Background] Nguyen HQ, Vallejo JD, Macias M, Shiffman MG, Rosen R, Mowry V, Omotunde O, Hong B, Liu IA, Borson S. A mixed-methods evaluation of home-based primary care in dementia within an integrated system. J Am Geriatr Soc. 2022 Apr;70(4):1136-1146. doi: 10.1111/jgs.17627. Epub 2021 Dec 22. PMID 34936090
- [Background] Sorensen S, Conwell Y. Issues in dementia caregiving: effects on mental and physical health, intervention strategies, and research needs. Am J Geriatr Psychiatry. 2011 Jun;19(6):491-6. doi: 10.1097/JGP.0b013e31821c0e6e. No abstract available. PMID 21502853
- [Background] Brodaty H, Donkin M. Family caregivers of people with dementia. Dialogues Clin Neurosci. 2009;11(2):217-28. doi: 10.31887/DCNS.2009.11.2/hbrodaty. PMID 19585957
- [Background] Chiao CY, Wu HS, Hsiao CY. Caregiver burden for informal caregivers of patients with dementia: A systematic review. Int Nurs Rev. 2015 Sep;62(3):340-50. doi: 10.1111/inr.12194. Epub 2015 Jun 8. PMID 26058542
- [Background] Li L, Wister AV, Mitchell B. Social Isolation Among Spousal and Adult-Child Caregivers: Findings From the Canadian Longitudinal Study on Aging. J Gerontol B Psychol Sci Soc Sci. 2021 Aug 13;76(7):1415-1429. doi: 10.1093/geronb/gbaa197. PMID 33170276
- [Background] Schulz R, O'Brien AT, Bookwala J, Fleissner K. Psychiatric and physical morbidity effects of dementia caregiving: prevalence, correlates, and causes. Gerontologist. 1995 Dec;35(6):771-91. doi: 10.1093/geront/35.6.771. PMID 8557205
- [Background] Heintz H, Monette P, Epstein-Lubow G, Smith L, Rowlett S, Forester BP. Emerging Collaborative Care Models for Dementia Care in the Primary Care Setting: A Narrative Review. Am J Geriatr Psychiatry. 2020 Mar;28(3):320-330. doi: 10.1016/j.jagp.2019.07.015. Epub 2019 Aug 2. PMID 31466897
- [Background] Tanner JA, Black BS, Johnston D, Hess E, Leoutsakos JM, Gitlin LN, Rabins PV, Lyketsos CG, Samus QM. A randomized controlled trial of a community-based dementia care coordination intervention: effects of MIND at Home on caregiver outcomes. Am J Geriatr Psychiatry. 2015 Apr;23(4):391-402. doi: 10.1016/j.jagp.2014.08.002. Epub 2014 Aug 13. PMID 25260557
- [Background] Possin KL, Merrilees JJ, Dulaney S, Bonasera SJ, Chiong W, Lee K, Hooper SM, Allen IE, Braley T, Bernstein A, Rosa TD, Harrison K, Begert-Hellings H, Kornak J, Kahn JG, Naasan G, Lanata S, Clark AM, Chodos A, Gearhart R, Ritchie C, Miller BL. Effect of Collaborative Dementia Care via Telephone and Internet on Quality of Life, Caregiver Well-being, and Health Care Use: The Care Ecosystem Randomized Clinical Trial. JAMA Intern Med. 2019 Dec 1;179(12):1658-1667. doi: 10.1001/jamainternmed.2019.4101. PMID 31566651
- [Background] Arora S, Thornton K, Murata G, Deming P, Kalishman S, Dion D, Parish B, Burke T, Pak W, Dunkelberg J, Kistin M, Brown J, Jenkusky S, Komaromy M, Qualls C. Outcomes of treatment for hepatitis C virus infection by primary care providers. N Engl J Med. 2011 Jun 9;364(23):2199-207. doi: 10.1056/NEJMoa1009370. Epub 2011 Jun 1. PMID 21631316
- [Background] Stammen LA, Stalmeijer RE, Paternotte E, Oudkerk Pool A, Driessen EW, Scheele F, Stassen LP. Training Physicians to Provide High-Value, Cost-Conscious Care: A Systematic Review. JAMA. 2015 Dec 8;314(22):2384-400. doi: 10.1001/jama.2015.16353. PMID 26647260
- [Background] Ramsey AT, Proctor EK, Chambers DA, Garbutt JM, Malone S, Powderly WG, Bierut LJ. Designing for Accelerated Translation (DART) of Emerging Innovations in Health. J Clin Transl Sci. 2019 Jun;3(2-3):53-58. doi: 10.1017/cts.2019.386. Epub 2019 Jul 30. PMID 31528365
- [Background] Aarons GA, Hurlburt M, Horwitz SM. Advancing a conceptual model of evidence-based practice implementation in public service sectors. Adm Policy Ment Health. 2011 Jan;38(1):4-23. doi: 10.1007/s10488-010-0327-7. PMID 21197565
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Shih WJ, Ohman-Strickland PA, Lin Y. Analysis of pilot and early phase studies with small sample sizes. Stat Med. 2004 Jun 30;23(12):1827-42. doi: 10.1002/sim.1807. PMID 15195318
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Krueger, RA, Casey MA. Focus groups: a practical guide for applied research. Thousand Oaks, CA: SAGE Publications, Inc.; 2000.
- [Background] Summit virtual meeting series: 2020 national research summit on care, services, and supports for persons with dementia and their caregivers. [Internet]. National Institute on Aging. 2020 [cited 2022 Apr 25]; Available from: https://www.nia.nih.gov/2020-dementia-care-summit
- [Background] Medical care at home comes of age. [Internet]. California Health Care Foundation. 2021[cited 2022 Apr 25]; Available from: https://www.chcf.org/publication/medical-care-home-comes-age/
- [Background] Lucero KS. Net Promoter Score (NPS): What Does Net Promoter Score Offer in the Evaluation of Continuing Medical Education? J Eur CME. 2022 Nov 29;11(1):2152941. doi: 10.1080/21614083.2022.2152941. eCollection 2022. PMID 36465493
- [Background] Torisson G, Stavenow L, Minthon L, Londos E. Reliability, validity and clinical correlates of the Quality of Life in Alzheimer's disease (QoL-AD) scale in medical inpatients. Health Qual Life Outcomes. 2016 Jun 14;14:90. doi: 10.1186/s12955-016-0493-8. PMID 27301257
- [Background] Gramling R, Stanek S, Ladwig S, Gajary-Coots E, Cimino J, Anderson W, Norton SA; AAHPM Research Committee Writing Group; Aslakson RA, Ast K, Elk R, Garner KK, Gramling R, Grudzen C, Kamal AH, Lamba S, LeBlanc TW, Rhodes RL, Roeland E, Schulman-Green D, Unroe KT. Feeling Heard and Understood: A Patient-Reported Quality Measure for the Inpatient Palliative Care Setting. J Pain Symptom Manage. 2016 Feb;51(2):150-4. doi: 10.1016/j.jpainsymman.2015.10.018. Epub 2015 Nov 17. PMID 26596879
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Derived] Ritchie C, Leff B, Sy M, Thacker A, Donelan K, Forester B, Sheehan OC; Dementia Care Quality at Home Writing Group. Feasibility and Acceptability of a Clinician-Caregiver Co-Designed Dementia Care Intervention for Home-Based Primary Care. J Am Geriatr Soc. 2025 Dec;73(12):3849-3858. doi: 10.1111/jgs.70112. Epub 2025 Sep 21. PMID 40976934
- [Derived] Sy M, Thacker A, Sheehan OC, Leff B, Ritchie CS. Caring for caregivers and persons living with dementia under home-based primary care: protocol for an interventional clinical trial. Pilot Feasibility Stud. 2024 Feb 9;10(1):28. doi: 10.1186/s40814-024-01455-x. PMID 38336779

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dementia Care Quality at Home
Started (50 caregivers received the Dementia Care Quality at Home Intervention) | 50
Caregivers Enrolled | 50
Practice Personnel Enrolled | 21
Completed | 39
Not Completed | 11

BASELINE CHARACTERISTICS:
Population: Only the caregivers people living with dementia were enrolled in the study. The baseline data just reflects that of the caregiver or their reported measure of their care recipient living with dementia.
Arm/Group | Dementia Care Quality at Home
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 13
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50
Role of Caregiver [Count of Participants; unit: Participants]
  Adult Child | 27
  Facility Caregiver | 9
  Spouse/Partner | 7
  Niece | 3
  Private Paid Caregiver | 3
  Sibling | 1
Hours Spent Caregiving per week [Mean (Standard Deviation); unit: hours per week] | 88 (60)
Quality of Life in Alzheimer's Disease [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life in Alzheimer's Disease (QoL-AD) questionnaire is scored by summing responses to its 13 items, each rated on a 4-point Likert scale from 1 (poor) to 4 (excellent), to yield a total score between 13 and 52. Higher scores reflect better perceived quality of life. The total score can be interpreted across the continuum of quality of life, with lower scores indicating poorer quality of life and higher scores indicating better quality of life.
  This measure is a caregiver reported measure on behalf of their care recipient living with dementia
  units on a scale | 26 (5)
The Neuropsychiatric Inventory Questionnaire: Severity Score [Mean (Standard Deviation); unit: units on a scale] — The Neuropsychiatric Inventory Questionnaire (NPI-Q) severity score is calculated by summing responses to its 12 items, each rated on a 3-point scale from 1 (mild) to 3 (severe), to yield a total score between 0 and 36. Higher scores indicate greater severity of neuropsychiatric symptoms. The total score reflects the overall burden of symptom severity, with lower scores indicating minimal or absent symptoms and higher scores reflecting more severe symptomatology.
  units on a scale | 10 (7)
The Neuropsychiatric Inventory Questionnaire: Distress Score [Mean (Standard Deviation); unit: units on a scale] — The Neuropsychiatric Inventory Questionnaire (NPI-Q) distress score is calculated by summing caregiver ratings of the distress caused by each of the 12 symptoms, scored on a 6-point scale from 0 (not at all distressing) to 5 (extremely distressing), to yield a total score between 0 and 60. Higher scores indicate greater caregiver distress associated with patients' neuropsychiatric symptoms. The total score reflects the overall emotional and psychological burden on caregivers, with lower scores suggesting minimal distress and higher scores indicating more severe caregiver distress.
  units on a scale | 14 (12)
Zarit Burden Interview Score [Mean (Standard Deviation); unit: units on a scale] — The Zarit Burden Interview (ZBI) is scored by summing responses to its 22 items on a 5-point Likert scale, from 0 (not at all) to 4 (nearly always), to yield a total score between 0 and 88, with higher scores indicating greater caregiver burden. The total score is then interpreted within defined ranges: 0-21 for little or no burden, 21-40 for mild to moderate burden, 41-60 for moderate to severe burden, and 61-88 for severe burden.
  units on a scale | 16 (11)
Patient Health Questionnaire 8 Item Score [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire-8 (PHQ-8) is scored by summing responses to its 8 items, each rated on a 4-point scale from 0 (not at all) to 3 (nearly every day), to yield a total score between 0 and 24. Higher scores indicate greater depressive symptom severity. The total score is typically interpreted within defined ranges: 0-4 for none or minimal depression, 5-9 for mild depression, 10-14 for moderate depression, 15-19 for moderately severe depression, and 20-24 for severe depression.
  units on a scale | 5 (4)
Care Ecosystem Caregiver Self-Efficacy Score [Mean (Standard Deviation); unit: units on a scale] — Caregivers rate their self-efficacy on a 5-point scale of whether they strongly agree, agree, neutral, disagree, or strongly disagree to 4 items. (minimum score of 4, maximum score of 20, with higher score indicating higher self-efficacy)
  I know where to get the services I need.
  I have people I can turn to when I need help with my problems.
  I feel confident that I can manage future caregiving challenges.
  I feel confident that I can manage (name of the person with dementia)'s changes in behavior.
  units on a scale | 8 (3)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility for the Caregiver to Engage With and Complete Baseline Assessments.
Description: The percentage of identified caregivers who complete baseline assessments.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Dementia Care Quality at Home
Number analyzed (Participants) | 50
Participants | 50

2. Primary Outcome: Feasibility for the Caregiver to Access Educational Materials and Community Resources.
Description: Percent of caregivers will report using 1 or more materials provided by the practice.
Time Frame: Post-intervention (6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Dementia Care Quality at Home
Number analyzed (Participants) | 50
Participants | 50

3. Primary Outcome: Feasibility for the Practice of Identifying Potential Patients/Caregivers
Description: Ability of practice to generate list of their patients living with dementia using a questionnaire to the practice
Time Frame: Baseline
Population: % of practice staff that "agree" or "strongly agree" that "it was easy for our practice to generate a list of persons living with dementia"
Measure: Count of Participants; unit: Participants
Groups:
- Dementia Care Quality at Home: Practice personnel across two sites implementing the Dementia Care Quality at Home intervention.
Arm/Group | Dementia Care Quality at Home
Number analyzed (Participants) | 21
Participants | 18

4. Primary Outcome: Feasibility for the Practice of Assessing Eligible Patient/Caregiver Dyads.
Description: Ability of practice to identify eligible patient/caregiver dyads (e.g., caregiver experiencing burden or distress).
Time Frame: Baseline
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Dementia Care Quality at Home
Number analyzed (Participants) | 21
Participants | 18

5. Primary Outcome: Feasibility for the Practice to Use Baseline Assessments.
Description: Percent of practice personnel who conduct assessments that rate assessments as feasible to use
Time Frame: Post-intervention (6 months)
Population: > 75% practice personnel who conduct assessments will "agree" or "strongly agree" that assessments were feasible to use
Measure: Count of Participants; unit: Participants
Arm/Group | Dementia Care Quality at Home
Number analyzed (Participants) | 21
Participants | 18

6. Primary Outcome: Feasibility for the Practice to Complete Baseline Assessments
Description: The percent of audited assessments that are completed.
Time Frame: Post-intervention (6 months)
Population: 75% of audited assessments will be completed
Measure: Count of Units; unit: assessments
Units Other Than Participants: assessments
Arm/Group | Dementia Care Quality at Home
Number analyzed (Participants) | 10
Number analyzed (assessments) | 10
assessments | 7

7. Secondary Outcome: Feasibility for the Practice of Recruiting Patient/Caregiver Dyads
Description: Percentage of eligible dyads who enroll.
Time Frame: Pre-intervention
Population: The number of participants analyzed is greater than 50 as 80 is the number of dyads that were eligible for the study
Measure: Count of Participants; unit: Participants
Arm/Group | Dementia Care Quality at Home
Number analyzed (Participants) | 80
Participants | 50

8. Secondary Outcome: Patient Quality of Life
Description: Quality of Life in Alzheimer's Disease. The QoL-AD is comprised of 13 items (physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores, ability to do things for fun, money and life as a whole). Response options include 1(poor), 2(fair), 3(good) and 4 (excellent), for a total score of 13-52, with higher scores indicating better QoL.
Time Frame: Pre-Intervention (baseline) and post-intervention (6 months)
Population: Quality of Life in Alzheimer's Disease score Pre and Post-Intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dementia Care Quality at Home
Number analyzed (Participants) | 50
score on a scale
  QoL-AD Pre-Intervention | 25.5 [24.2 to 26.8]
  QoL-AD Post-Intervention: number analyzed (Participants) | 39
  QoL-AD Post-Intervention | 28.5 [26.6 to 30.4]

9. Secondary Outcome: Heard and Understood
Description: A one-item measure of caregivers who report that they felt heard and understood by the practice.
Time Frame: Post Intervention (6 months)
Population: % of caregivers who report that they felt heard and understood "quite a bit" or "completely" by the practice
Measure: Count of Participants; unit: Participants
Arm/Group | Dementia Care Quality at Home
Number analyzed (Participants) | 39
Participants | 37

10. Secondary Outcome: Caregivers - Net Promoter Score of Intervention
Description: The single question - "How likely are you to recommend X to a friend [or colleague]?" is rated from 0 - Not at all likely to 10 - Extremely likely.
Time Frame: Post-intervention (6 months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dementia Care Quality at Home
Number analyzed (Participants) | 39
score on a scale | 8.8 [8.2 to 9.4]

11. Secondary Outcome: Feasibility for the Practice to Use Care Modules.
Description: The percentage that rates modules as feasible to use. The percentage of practice personnel who complete the modules that rate the modules as feasible to use
Time Frame: Post-intervention (6 months)
Population: > 75% practice personnel who complete the modules will rate the modules as "feasible" or "very feasible" to use > 50% of audited modules will be completed
Measure: Count of Participants; unit: Participants
Arm/Group | Dementia Care Quality at Home
Number analyzed (Participants) | 21
Participants | 18

12. Secondary Outcome: Feasibility for the Practice to Complete Care Modules
Description: Percent of audited modules that are completed.
Time Frame: Post Intervention (6-months)
Population: > 50% of audited modules will be completed
Measure: Count of Units; unit: modules
Units Other Than Participants: modules
Arm/Group | Dementia Care Quality at Home
Number analyzed (Participants) | 12
Number analyzed (modules) | 12
modules | 11

13. Secondary Outcome: Feasibility for the Practice of Clinicians to Engage With the Tele-video Case Conference.
Description: % of case conferences conducted with at least one staff member present from each site
Time Frame: Post-intervention (6 months)
Measure: Count of Units; unit: case conferences attended
Units Other Than Participants: case conferences attended
Arm/Group | Dementia Care Quality at Home
Number analyzed (Participants) | 21
Number analyzed (case conferences attended) | 25
case conferences attended | 25

14. Secondary Outcome: Acceptability of the Intervention to Caregivers to Participate in the Intervention.
Description: Percent of caregivers invited to participate who agree to participate in the intervention.
Time Frame: Pre-intervention (baseline)
Population: The number of participants analyzed is greater than 50, as 80 is the number of dyads that were eligible for the study and invited to participate, 50 out of 80 enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Dementia Care Quality at Home
Number analyzed (Participants) | 80
Participants | 50

15. Secondary Outcome: Feasibility for the Practice of Percent of Racial and Ethnic Minorities Recruited.
Description: Percentage of eligible dyads who enroll who are racial and ethnic minorities.
Time Frame: Pre-intervention (baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Dementia Care Quality at Home
Number analyzed (Participants) | 50
Participants | 26

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline to the end of data collection, over 6 months.
Description: The definition of an adverse event or serious adverse event do not differ from the CT.gov definitions
Groups:
- Dementia Care Quality at Home Caregivers: Caregivers across two HBPC practices receive the Dementia Care Quality at Home intervention.
- Dementia Care Quality at Home Practice Personnel: Practice personnel implementing the Dementia Care Quality at Home Intervention
Arm/Group | Dementia Care Quality at Home Caregivers | Dementia Care Quality at Home Practice Personnel
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/21
Other Adverse Events (participants affected / at risk) | 0/50 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT05849259/Prot_SAP_000.pdf